CLINICAL TRIAL: NCT00770640
Title: Comparison of the Effects of Pioglitazone vs. Placebo When Given in Addition to Standard Insulin Treatment in Patients With Type 2 Diabetes Mellitus and Renal Failure
Brief Title: Efficacy of Pioglitazone and Insulin in Treating Subjects With Type 2 Diabetes Mellitus and Renal Failure.
Acronym: PIOren
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Takeda (Industry)
Responsible Party: Medical Director, Takeda Pharma GmbH, Aachen (Germany)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ATS K029; 2007-006744-21 (EudraCT Number); DE-PIO-029 (Other: Takeda ID); U1111-1114-1645 (Registry Identifier: WHO)
Record Dates: First submitted 2008-10-09; First posted 2008-10-10 (Estimated); Last update posted 2010-09-01 (Estimated); Status verified 2010-08

CONDITIONS: Diabetes Mellitus
Keywords: Glucose Metabolism Disorder; Dysmetabolic Syndrome; Type II Diabetes; Diabetes Mellitus, Lipoatrophic; Dyslipidemia; Drug Therapy
MeSH Terms: conditions — Diabetes Mellitus; Glucose Metabolism Disorders; Diabetes Mellitus, Type 2; Diabetes Mellitus, Lipoatrophic; Dyslipidemias | interventions — Pioglitazone; Insulin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Pioglitazone 30mg QD (Experimental): (and variable insulin therapy)
  Interventions: Drug: Pioglitazone and insulin
- Placebo QD (Placebo Comparator): (and variable insulin therapy)
  Interventions: Drug: Insulin

INTERVENTIONS:
Drug: Pioglitazone and insulin — Pioglitazone 30 mg, tablets, orally, once daily and variable insulin therapy for up to 24 weeks.
  Other Names: ACTOS®; AD-4833
  Arms: Pioglitazone 30mg QD
Drug: Insulin — Pioglitazone placebo-matching tablets, orally, once daily and variable insulin therapy for up to 24 weeks.
  Arms: Placebo QD

SUMMARY:
The purpose of this study is to determine the metabolic and cardiovascular effects of pioglitazone, once daily (QD), and insulin combination therapy in subjects with Type 2 Diabetes and Renal Failure.

DETAILED DESCRIPTION:
Patients with type 2 diabetes mellitus and clinically significant kidney disease presenting with contra-indications for metformin and sulfonylurea drugs are usually treated with insulin therapy only. While the prolonged pharmacokinetic insulin profile due to delayed renal insulin elimination already is a hurdle for a successful therapy, impaired kidney function results in increased oxidative stress and cardiovascular risk, especially in patients requiring dialysis. Several potential mechanisms may explain this increased cardiovascular risk, and one, frequent finding is coexistence of several other independent cardiovascular risk factors including dyslipidemia, hypertension and smoking. In addition, impaired kidney function is associated with elevated markers of inflammation and other putative risk factors for cardiovascular events.

The focus of this study is to investigate whether pioglitazone may help improve overall metabolic and cardiovascular risks in patients with end stage renal disease, and if pioglitazone can potentially exert positive effects on kidney function in patients with renal failure requiring dialysis.

The duration of treatment for patients completing the study is approximately 26 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Has Type 2 Diabetes Mellitus, and is a patient on insulin treatment for at least 3 months.
* Has a body mass index less than 36 kg/m²
* Has a glycosylated hemoglobin level greater than or equal to 6.0% and less than 10%.
* Patient is on hemo-dialysis with or without residual excretion
* An insulin dose greater than 20 IE/day

Exclusion Criteria:

* Has a history of type 1 diabetes.
* Has acute infections.
* History of hypersensitivity to the study drugs or to drugs with similar chemical structures.
* History of severe or multiple allergies.
* Has a progressive fatal disease other than kidney failure.
* Has a history of drug or alcohol abuse within the last 5 years.
* A history of significant cardiovascular (e.g. Coronary heart failure based on New York Heart Association stage III - IV), respiratory, gastrointestinal, hepatic (e.g. alanine aminotransferase greater than 2.5 times the normal reference range) or hematological disease.
* History of primary hyperaldosteronism
* Acute myocardial infarction, open heart surgery or cerebral event (stroke/transient ischemic attack) within the last year prior to study start.
* Any further antidiabetic treatment except pioglitazone and insulin.
* History of macular edema.
* Is required to take or intends to continue taking any disallowed medication, any prescription medication, herbal treatment or over-the counter medication that may interfere with evaluation of the study medication, including:

  * Treatment with any other investigational drug within 3 months before trial entry.
  * Treatment with steroids within 3 months before trial entry.
  * Treatment with thiazolidinediones within the past 3 months.
  * If statin therapy applicable: Change of medication within the last 4 weeks.
  * Pre-treatment with gemfibrozil within the last 12 weeks.
  * Pre-treatment with rifampicin within the last 12 weeks.
* Has uncontrolled unstable angina.

Ages: 30 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2008-08; Primary Completion 2010-06 (Actual); Study Completion 2010-06 (Actual)

PRIMARY OUTCOMES:
Change of total daily Insulin Dose. | Week 24 or Final Visit.

SECONDARY OUTCOMES:
Individual insulin doses to assess the number of patients with insulin reduction of greater than or equal to 30%. | Weeks 12 and 24 or Final Visit.
Change from Baseline in Glycosylated Hemoglobin. | Weeks 12 and 24 or Final Visit.
Change from Baseline in Glucose. | Weeks 12 and 24 or Final Visit.
Change from Baseline in Insulin. | Weeks 12 and 24 or Final Visit.
Change from Baseline in C-peptide. | Weeks 12 and 24 or Final Visit.
Change from Baseline in Intact Proinsulin. | Weeks 12 and 24 or Final Visit.
Change from Baseline in Adiponectin. | Weeks 12 and 24 or Final Visit.
Change from Baseline in Angiotensin. | Weeks 12 and 24 or Final Visit.
Change from Baseline in Relaxin. | Weeks 12 and 24 or Final Visit.
Change from Baseline in fetuin A. | Weeks 12 and 24 or Final Visit.
Change from Baseline in Carbonyl Protein. | Weeks 12 and 24 or Final Visit.
Change from Baseline in Myeloperoxidase. | Weeks 12 and 24 or Final Visit.
Change from Baseline in Matrix-Gla Protein. | Weeks 12 and 24 or Final Visit.
Change from Baseline in High Sensitivity C-reactive Protein. | Weeks 12 and 24 or Final Visit.
Change from Baseline in Cholesterol. | Weeks 12 and 24 or Final Visit.
Change from Baseline in High-Density Lipoprotein. | Weeks 12 and 24 or Final Visit.
Change from Baseline in Low-Density Lipoprotein. | Weeks 12 and 24 or Final Visit.
Change from Baseline in Oxidized Low-Density Lipoprotein. | Weeks 12 and 24 or Final Visit.
Change from Baseline in Triglycerides. | Weeks 12 and 24 or Final Visit.
Change from Baseline in Matrix Metalloproteinase -9. | Weeks 12 and 24 or Final Visit.
Change from Baseline in Monocyte Chemoattractant Protein -1. | Weeks 12 and 24 or Final Visit.
Change from Baseline in E-selectin. | Weeks 12 and 24 or Final Visit.
Pioglitazone in serum. | Week 12.
Change from Baseline in intact Parathyroid Hormone. | Weeks 12 and 24 or Final Visit.

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Takeda Pharma GmbH, Aachen (Germany)
Locations (9):
- Germany (9):
  - Schwetzingen, Baden-Wurttemberg
  - Wiesbaden, Hesse
  - Bottrop, North Rhine-Westphalia
  - Düsseldorf, North Rhine-Westphalia
  - Lüdenscheid, North Rhine-Westphalia
  - Solingen, North Rhine-Westphalia
  - Alzey, Rhineland-Palatinate
  - Ingelheim, Rhineland-Palatinate
  - Mainz, Rhineland-Palatinate

REFERENCES:
- See also: ACTOS® Package Insert — http://general.takedapharm.com/content/file/pi.pdf?applicationcode=ab2d7112-8eb3-465a-8fda-35018a9eafb0&fileTypeCode=ACTOSPI